# **Official Study Title**

Biomarker Studies to Predict Treatment Outcomes of Enfortumab Vedotin in Advanced Urothelial Carcinoma

ClinicalTrials.gov Identifier (NCT Number): Pending Assignment

Document Date: June 19, 2025

### **Confidentiality Notice:**

This document is intended for use in the ClinicalTrials.gov registration and results reporting process only. It does not contain any personal identifiers of study participants.

### 1. Official Study Title

Biomarker Studies to Predict Treatment Outcomes of Enfortumab Vedotin in Advanced Urothelial Carcinoma

### 2. Background and Rationale

Advanced urothelial carcinoma (aUC) remains a highly fatal malignancy, with limited durable responses to first-line platinum-based chemotherapy. Enfortumab vedotin (EV), a nectin-4-targeting antibody-drug conjugate, has shown promising efficacy in aUC patients, both in the first-line setting when combined with pembrolizumab and in later-line setting when used as monotherapy (EV/EVP). However, despite its clinical success, the occurrence of significant toxicities and high treatment costs highlight the need for predictive biomarkers to optimize treatment outcomes and mitigate adverse effects. Nectin-4, as the target of EV, along with ADAM10/17, enzymes responsible for nectin-4 shedding, and soluble nectin-4 (sNectin-4), have emerged as potential biomarkers for predicting EV treatment outcomes.

### 3. Objectives

### 3-1. Primary Objective

(1) To investigate the correlation between membranous nectin-4 (mNectin-4) expression and treatment outcomes in patients with aUC receiving EV/EV-P.

#### 3-2. Secondary Objectives

- (1) To evaluate the association between ADAM10/17 expression and treatment outcomes of EV/EVP in aUC.
- (2) To examine the relationship between sNectin-4 levels and treatment efficacy of EV/EVP in aUC patients.

#### 3-3. Exploratory Objective

(1) To assess whether mNectin-4, ADAM10/17, and sNectin-4 can serve as predictive biomarkers for EV/EVP in aUC patients.

### 4. Study Design

- 4-1. Study Type: Observational
- 4-2. Study Design: Prospective cohort study
- 4-3. **Study Center**: Single-center (National Taiwan University Hospital, NTUH); may expand to multi-center in the future
- 4-4. Enrollment Method: Consecutive enrollment of eligible patients
- 4-5. **Study Period**: April 1, 2025 to December 31, 2029
- 4-6. **Estimated Sample Size**: 100 patients receiving EV/EVP, plus 100 patients treated with platinum-based chemotherapy as a comparator cohort

### 5. Study Population

### 5-1. Inclusion Criteria

- (1) Histologically confirmed diagnosis of advanced aUC, including bladder cancer or upper tract urothelial carcinoma
- (2) Age  $\geq$  20 years
- (3) Received EV/EVP or first-line platinum-based chemotherapy at NTUH

- (4) Availability of archival formalin-fixed paraffin-embedded (FFPE) tumor tissue for biomarker analysis
- (5) Willingness to provide serum samples at predefined time points
- (6) Ability to provide written informed consent

#### 5-2. Exclusion Criteria

- (1) Patients who have received prior investigational agents targeting nectin-4
- (2) Inadequate tissue samples or insufficient serum collection
- (3) Concurrent participation in another interventional clinical trial
- (4) Any condition that, in the investigator's judgment, would compromise the patient's safety or compliance with study procedures

#### 5-3. Sampling Method

(1) Consecutive enrollment of eligible patients meeting the inclusion criteria

#### 5-4. Estimated Sample Size

- (1) 100 patients treated with EV/EVP
- (2) 100 patients treated with first-line platinum-based chemotherapy (for comparative biomarker analysis)

### 6. Study Groups/Cohorts

### 6-1. Group 1: EV Therapy Cohort

- (1) Population: Patients with aUC receiving EV/EVP at NTUH
- (2) Treatment: Standard EV-based regimen (monotherapy or in combination with pembrolizumab)
- (3) Biospecimen Collection:
  - Archival tumor tissue for immunohistochemistry (IHC) analysis of mNectin-4 and ADAM10/17 expression
  - o Serum samples collected at predefined time points for sNectin-4 quantification via ELISA

(4) Clinical Data Collection: Demographics, disease characteristics, treatment details, response assessments (RECIST), progression-free survival, overall survival, and adverse events

#### 6-2. Group 2: Chemotherapy Cohort (Comparator Cohort)

- (1) Population: Patients with aUC who received first-line platinum-based chemotherapy at NTUH during the same enrollment period
- (2) Treatment: Standard first-line cisplatin- or carboplatin-based chemotherapy
- (3) Biospecimen Collection:
  - o Archival tumor tissue for IHC analysis of mNectin-4 and ADAM10/17
  - o Serum samples for sNectin-4 quantification
- (4) Clinical Data Collection: As per EV therapy cohort, for comparative analysis

### 7. Endpoints / Outcome Measures

### 7-1. Primary Outcome Measure

(1) Objective Response Rate (ORR): Proportion of patients achieving complete or partial tumor response according to RECIST 1.1 criteria after enfortumab vedotin treatment. Time Frame: Up to 12 months after treatment initiation

### 7-2. Secondary Outcome Measure

- (1) Progression-Free Survival (PFS): Time from treatment start to disease progression or death from any cause. Time Frame: Up to 24 months
- (2) Overall Survival (OS): Time from treatment initiation to death from any cause. Time Frame: Up to 36 months
- (3) Treatment-Related Adverse Events: Incidence and severity of adverse events graded by CTCAE v5.0

during treatment. Time Frame: Throughout treatment duration

(4) Correlation of Biomarker Expression with Treatment Outcomes: Association between mNectin-4, ADAM10/17 expression, serum sNectin-4 levels, and clinical outcomes. Time Frame: Assessed at baseline and during follow-up

### 8. Methods / Assessments

#### 8-1. Sample Collection

### (1) Tumor Tissue:

- Archival formalin-fixed paraffin-embedded (FFPE) tumor specimens will be retrieved from diagnostic pathology samples.
- o Tumor samples will be analyzed for mNectin-4 and ADAM10/17 expression by IHC.

### (2) Serum Samples:

- Blood samples will be collected at predefined time points: before the initiation of systemic therapies/at first radiographic response assessment (approximately week 6–8)/t disease progression or end of treatment
- o Serum will be isolated and stored at -80°C for subsequent analysis of sNectin-4 by ELISA.

#### 8-2. Biomarker Analysis

#### (1) IHC:

- o FFPE tissue sections will be stained for nectin-4 and ADAM10/17 using validated antibodies.
- Expression will be semi-quantitatively scored based on H-score and/or staining intensity and proportion.

#### (2) Enzyme-Linked Immunosorbent Assay (ELISA):

 Serum sNectin-4 levels will be quantified using a commercially available ELISA kit following manufacturer's instructions.

#### 8-3. Statistical Analysis

- (1) Descriptive statistics will be used to summarize patient characteristics and biomarker distributions.
- (2) Group comparisons:
  - Mann–Whitney U test or t-test for continuous variables
  - o Chi-square or Fisher's exact test for categorical variables
- (3) Survival analysis:
  - Kaplan–Meier method for estimating PFS and OS
  - Log-rank test for between-group comparisons
- (4) Multivariable analysis:
  - o Cox proportional hazards model to assess the independent association of biomarkers with survival outcomes
  - Logistic regression for associations with objective response

### 9. Ethics / Regulatory Compliance

9-1. The study protocol has been reviewed and approved by the Research Ethics Committee E of **National Taiwan University Hospital.** 

IRB Approval Number: 202502065RINE

Approval Date: 2025-03-19

- 9-2. This study will be conducted in accordance with the principles of the Declaration of Helsinki, ICH Good Clinical Practice (GCP) guidelines, and applicable local regulatory requirements.
- 9-3. Informed consent will be obtained from all participants before enrollment. The consent process will include information on study purpose, procedures, risks, benefits, data confidentiality, and the

voluntary nature of participation.

### 9-4. Confidentiality and data protection:

- All personal identifying information will be coded and stored securely in password-protected databases.
- o Only authorized study personnel will have access to identifiable data.
- o Samples will be labeled with de-identified study codes.
- o Data will be reported in aggregate to prevent the identification of individual participants.

## **10. Study Timeline**

10-1. Planned Study Start Date: April 1, 2025

10-2. Planned Study End Date (Final Data Collection): December 31, 2029

10-3. Primary Completion Date: September 30, 2029

10-4. Study Completion Date: December 31, 2029